CLINICAL TRIAL: NCT07182578
Title: Programming Aquatic Therapy for POTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, Dominguez Hills (Other)
Responsible Party: Principal Investigator, EvaRose Celeste, Principal Investivator, California State University, Dominguez Hills
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2025-162
Record Dates: First submitted 2025-09-10; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS)
Keywords: Aquatic Therapy; Occupational therapy; POTS; Postural Orthostatic Tachycardia Syndrome; Dysautonomia; Rehabilitation; Hydrotherapy
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Autonomic Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquatic Occupational Therapy Intervention (Experimental): All participants will participate in the aquatic occupational therapy arm. The aquatic occupational therapy intervention is divided into three progressive months:
  Month 1: Breathing techniques, proprioception, balance, and vestibular activities.
  Easy breathing and balancing moves Example: Belly breathing, water walking, toe lifts, mountain aqua yoga pose Month 2: Strength and endurance training Building strength and ability to exercise longer Example: Water marching, core exercises using dumbbells or paddles Month 3: Advanced strengthening and endurance tasks with integrated cognitive, balance, and dual-task challenges.
  Harder exercises and doing two things at once, like thinking and moving together Example: Dumbbell exercises while playing a word association game
  Interventions: Other: Aquatic Occupational Therapy

INTERVENTIONS:
Other: Aquatic Occupational Therapy — Aquatic Occupational Therapy sessions will be 60 minutes long, with 45 minutes spent in the pool. Sessions will include a gentle floating, stretching, or aqua yoga warm-up and an ai chi cooldown. Exercises in the first month will include a focus on balance, breathing, and sensory work. Exercises in the second month will focus on building strength and endurance, while the third month will combine all of the above with dual-task completion. Activities will be graded down (made less difficult) or graded up (made more challenging) according to individual participant needs.

SUMMARY:
The goal of this pilot study is to create, implement, and evaluate an aquatic therapy for Postural Orthostatic Tachycardia Syndrome (POTS) program feasibility and ability to improve quality of life as determined by reduced orthostatic tachycardia, reduced POTS symptoms, and improved quality of life measures.

The main questions it aims to answer are:

Does aquatic occupational therapy reduce orthostatic tachycardia and POTS symptoms? Does aquatic occupational therapy lead to higher quality of live measures for people with POTS? Is this aquatic occupational therapy program feasible for clinicians and people with POTS?

There is no comparison group for this pilot study.

Participants will complete:

An occupational Therapy evaluation before and after program completion (3 hours total) 30 minutes at home/remote 30 minutes on-site/in-person 30 minutes of individualized occupational therapy on land

Participate in 3 aquatic therapy sessions per week, 60 minutes each for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with POTS, Age 18-64, Participants must be English speaking, participants must obtain a physician permission letter* * The physician letter will only state that the participant is cleared to participate in aquatic therapy, it will not confirm or state what disease the individual has in the medical records or other HIPAA information.

Exclusion Criteria:

* Not diagnosed with POTS, Not between the ages of 18-64*, Epilepsym Bowel incontinence

  *The reason for the age requirement is because individuals:
* under 18 have different diagnostic criteria and mechanisms for POTS than the age range specified and may respond differently to treatment
* over age 65 have different mechanisms behind POTS than younger individuals, and frequently have health conditions or factors that can be difficult to differentiate from POTS symptoms/diagnosis and would require lab work and continuous physician involvement. POTS is less common in older adults.
* The typical age of onset for POTS is generally considered to be between the ages of 15-50 years of age
* For participant's safety, the researcher needs to be able to communicate with them in the aquatic setting. English is the researcher's only language and electronic translators are not accessible/usable in the pool setting.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life - Brief (WHOQOL-BREF) | From enrollment to the end of 12 weeks of aquatic occupational therapy intervention
  The WHOQOL-BREF is a 26-item questionnaire that will be completed digitally. It is scored by first assigning numerical values (1-5) to each response, with higher scores generally indicating a better quality of life. Then, raw domain scores are calculated by averaging the responses within each domain (Physical, Psychological, Social, and Environmental). Finally, these raw domain scores are transformed into scaled scores ranging from 0 to 100 by multiplying by 4. Higher scores on the 0-100 scale indicate a higher quality of life.
  The measure will be reported as a quality of life score.
The DePaul Symptom Questionnaire (Short Form) (DSQ-SF) | From enrollment to the end of 12 weeks of aquatic occupational therapy intervention.
  14-item-questionnaire which measures post-exertional malaise symptoms over the last 6 months. Each question requires two ratings, one for frequency (0 = none of the time and 4 = all of the time) and one for severity (0 = symptom not present and 4 = very severe). A frequency of at least 2 and a severity of at least 2 on any one of the 5 questions on the DSQ-SF subscale indicate that post exertional malaise is present. For each symptom, the frequency and severity scores are averaged, and then multiplied by 25 to create a composite score out of 100.
  The measure will be reported as a post exertional malaise score.
Composite Autonomic Symptom Score-31 | From enrollment to the end of 12 weeks of aquatic occupational therapy intervention.
  Measures neurodegenerative system symptoms through 31 patient-reported questions. Assessment is through six weighted domains: orthostatic intolerance [10 points]; vasomotor [6 points]; secretomotor [7 points]; gastrointestinal [28 points]; bladder [9 points] and pupillomotor [15 points]. A higher score indicates worse autonomic dysfunction. Simple yes or no questions are scored as 0 points for no and 1 point for yes. Questions about a specific site of symptoms or symptoms under specific circumstances are scored as 0 if not present and as 1 if present for each site or circumstance. All questions regarding the frequency of symptoms were scored as 0 points for rarely or never, 1 point for occasionally or sometimes, 2 points for frequently or "a lot of the time," and 3 points for almost always or constantly. All questions regarding the severity of symptoms were scored as 1 point for mild, 2 points for moderate, and 3 points for severe.
  The measure will be reported as a COMPASS score
Malmo POTS Scale (MAPS) | From enrollment to the end of 12 weeks of aquatic occupational therapy intervention
  This 12-item questionnaire assesses the specific POTS symptom burden over the past 3 months. Each question uses a visual analog scale from 0-10, with a maximum score of 120. A score of 42 or higher is considered indicative of POTS.
  The measure will be reported as a MAPS score.
ADLS, IADLS, and Vestibular Questionnaire | From enrollment to the end of 12 weeks of aquatic occupational therapy intervention
  This is a 26-item questionnaire that will be filled out digitally. 21 questions cover about to participate in occupations listed in the Occupational Therapy Practice Framework using a scale from 1-10, where 1 is unable to complete the task, 5 is able to complete task with moderate difficulty (noticeable symptoms and extra effort is required) 10 is no problems/symptoms completing the task. It also contains 5 vestibular related questions using a scale from 1-7, with 1 being not at all dizzy, 4 being moderately dizzy, and 7 being extremely dizzy. The measure will be reported as an AIVQ score.
Active Stand Test | From enrollment until the end of treatment at 12 weeks
  The patient will begin laying down in a relaxed and comfortable position. Blood pressure (BP) and heart rate (HR) are taken after 5 minutes. Next, the patient will be asked to stand promptly, and will have their BP and HR measured immediately. The therapist will note any comments like "feeling dizzy". The BP and HR will be taken again and documented after three minutes, and again after ten minutes of standing. If there is any event, such as severe dizziness, paleness, etc, the BP and HR will be taken and documented just before the patient sits down.
  The measure will be reported as the position, time, and the correlated heart rate and blood pressure.
Single leg stance test | From enrollment to the end of 12 weeks of aquatic occupational therapy intervention
  This test measures a person's ability to balance standing on one leg without assistance. The participant will stand on one leg with their hands on their hips while being timed. The test is repeated 3 times for each leg and averaged. The measure will be reported as time standing per leg.
Heart Rate | From enrollment to the end of treatment at 12 weeks
  Heart rate (HR) will be measured on land while the participant is laying down, sitting up, and standing. HR in the water will be taken while seated and standing. An aquatic HR maximum and HR zones will be calculated for each participant. This measure will be reported as a land-based and aquatic HR maximum.
Borg's rate of perceived exertion scale | From enrollment to the end of treatment at 12 weeks
  This scale is used to tell how tiring an activity feels. The scale ranges from 6 (no exertion at all), to 20 (maximal heaviness). This will be reported as the RPE score.

SECONDARY OUTCOMES:
The Stroop Test | From enrollment to the end of 12 weeks of aquatic occupational therapy intervention
  The Stroop Test is a measure of working memory and attention. A participant is asked to read words of various colors, say the color of the letters when they are the same, and when the colors don't match the words. They are timed and errors are tracked. This will be reported as the SCWT score.
Trail Making Test Parts A & B | From enrollment to the end of the intervention at 12 weeks
  The participant is given a paper with numbers and letters, and is instructed to connect the letters and numbers in order (1-A-2-B-3-C, etc.), as quickly as possible, without lifting the pend or pencil from the paper. Errors will be pointed out immediately and the participant is allowed to correct it, but the time it takes to correct is still included in the completion time for the task. This will be reported as the TMT-A and TMT-B scores.
Enrollment | From enrollment to the end of treatment at 12 weeks
  Total number of participants who complete the informed consent, evaluation session, and agree to participate in program according to schedule discussed with participant
Attrition Rate | From enrollment to the end of treatment at 12 weeks
  The number of enrolled participants who do not complete the program
Session attendance rate | From enrollment to the end of treatment at 12 weeks
  This will be calculated by the number of sessions attended out of the total number of sessions for the program.
Cost analysis | From enrollment to the end of treatment at 12 weeks
  This measure will include resource tracking and total costs divided by the number of completers.
Health utilization changes | From enrollment to the end of treatment at 12 weeks
  This will include a calculation of health utilization changes from before the program compared to after the program
Satisfaction Analysis | From enrollment to the end of treatment at 12 weeks
  Thematic analysis of open-ended feedback from participants and stakeholders will determine the most common themes and areas for improvement within the program.
Exercise self-efficacy | From enrollment to the end of treatment at 12 weeks
  Measure will be completed before the program and compared to the result after, leading to an ESE score.

CONTACTS AND LOCATIONS:
Overall Officials: EvaRose Celeste, OT Doctoral student, Principal Investigator — California State University, Dominguez Hills; Tracy Becerra-Culqui, PhD, MPH, BS OT, Study Chair — California State University, Dominguez Hills
Locations (1):
- California Aquatic Therapy & Wellness Center, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
The final dataset will include individual-level vaccination and demographic data, as well as other health characteristics. We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. We will share the final dataset under our own auspices and by our own determination based on review of a detailed research plan submitted by the requestor.